CLINICAL TRIAL: NCT06145698
Title: The Exploration of Novel Cross-frequency Protocol of Transcranial Alternating Current Stimulation in the Treatment of Methamphetamine Use Disorder: A Randomized Sham-controlled Study
Brief Title: Treatment Effect of Cross-frequency Transcranial Alternating Current Stimulation on the MUD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MZhao-014
Record Dates: First submitted 2023-10-24; First posted 2023-11-24 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-10

CONDITIONS: Amphetamine-Related Disorders
MeSH Terms: conditions — Amphetamine-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: theta-gamma tACS (Experimental): The study is investigating the use of transcranial alternating current stimulation (tACS). For the experimental arm, the stimulation is delivered at 2 milliamperes (mA) with the stimulation electrode over the left prefrontal cortex (F3) and left orbitofrontal cortex (Fp1) using the cross-frequency stimulation waveform theta-gamma.
  Interventions: Device: Cross-frequency transcranial alternating current stimulation via the Neuroelectrics Starstim 32 transcranial electric stimulation device
- Active-sham tACS (Sham Comparator): For the active sham stimulation, the stimulation is delivered for 12 seconds with the theta-gamma cross-frequency stimulation waveform and then returns to baseline. The stimulus parameter of the sham stimulation is designed to mimic the adaptive sensations experienced by the subject when receiving the real stimulation treatment settings, but no effective brain modulation will be produced, which assists with blinding the participant's assignment.
  Interventions: Device: Cross-frequency transcranial alternating current stimulation via the Neuroelectrics Starstim 32 transcranial electric stimulation device

INTERVENTIONS:
Device: Cross-frequency transcranial alternating current stimulation via the Neuroelectrics Starstim 32 transcranial electric stimulation device — Stimulation will be delivered via the Neuroelectrics Starstim 32 transcranial electric stimulation device, an investigational electrical non-invasive brain stimulation device that is being used for clinical and translational research.

SUMMARY:
The purpose of this research is to evaluate the efficacy of multiple sessions of theta-gamma cross-frequency transcranial alternating current stimulation in patients with methamphetamine (MA) use disorders.

DETAILED DESCRIPTION:
Previous evidence suggests that different aspects of cognitive function are associated with activities of distinct EEG frequency bands. Gamma oscillatory has been found in clinical studies to reflect the processing of rewards in patients with drug dependence, whereas medial prefrontal theta oscillatory characterizes prefrontal response inhibition capacity to downstream reward arousal. Interestingly, impaired response inhibition or impaired evaluation of rewards in patients with drug dependence have been found to correlate with the arousal of psychological craving and the emergence of relapse. Here we aim to find causal evidence supporting these previous correlational findings by applying cross-frequency transcranial alternating current stimulation (tACS) in the specific frequency bands (theta-gamma) previously shown to be addiction-relevant. In a randomized control clinical trial design, we stimulate subjects with either theta-gamma or sham tACS. Electroencephalography will be collected before and after each treatment session. Besides, the scale and behavior task data will also collected before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. In accordance with the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) for methamphetamine (MA) use disorders
2. Normal vision and hearing
3. Dextromanual
4. Use MA not less than 1 year, and the last of MA use no less than 3 months

Exclusion Criteria:

1. Have a disease that affects cognitive function such as a history of head injury, cerebrovascular disease, epilepsy, etc
2. Have cognitive-promoting drugs in the last 6 months
3. Other substance abuse or dependence in recent five years (except nicotine)
4. Meet the DSM-5 criteria for other mental disorders
5. Physical disease

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Change of Craving assessed by Visual Analog Scale | baseline，0-2 days after treatment，1 months after treatment, 3 months after treatment
  evaluate all participants' craving for for methamphetamine assessed by Visual Analog Scales (VAS). Score of VAS range from 0 to 10, and higher values represent high level of craving.

SECONDARY OUTCOMES:
Depression status assessed by Beck Depression Inventory (BDI) | baseline，0-2 days after treatment，1 months after treatment, 3 months after treatment
  The reduction rate in the Beck Depression Inventory (BDI) scores was calculated before and after the treatment to evaluate the rate of reduction in their levels of depression.
Anxiety status assessed by Beck Anxiety Inventory (BAI) | baseline，0-2 days after treatment，1 months after treatment, 3 months after treatment
  The reduction rate in the Beck Anxiety Inventory (BAI) scores was calculated before and after treatment to assess the rate of decrease in anxiety levels among MA dependents.
Sleep Quality Assessment | baseline，0-2 days after treatment，1 months after treatment, 3 months after treatment
  Sleep Quality is assessed by the scores of Insomnia Severity Index(ISI) and Pittsburgh Sleep Quality Index(PSQI).
Brain oscillations | baseline，within 30 minutes before and after each session of treatment
  Assessed by Resting EEG task under the electroencephalogram recording to extract alpha, beta, theta, and gamma band energy.
Reward learning | baseline，0-2 days after treatment, 3 months after treatment
  Learning rate and the sensitivity to rewards assessed by Monetary reinforcement learning task under the electroencephalogram recording, and the results will be derived from modeling.
Spatial working memory | baseline，0-2 days after treatment, 3 months after treatment
  Working memory capacity is assessed by Spatial working memory under the electroencephalogram recording. The indicator is the correctness and response time.

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhao, PhD, Study Director — Shanghai Mental Health Center
Locations (1):
- Wuhan Compulsory Rehabilitation Center, Wuhan, China